CLINICAL TRIAL: NCT07401888
Title: Milk Consumption On Cardiovascular Risk Factors In Metabolic Syndrome
Brief Title: A Study Of Milk Consumption In Metabolic Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joshua R. Smith, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 25-010619
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-fat diet first then Low-fat diet (Experimental)
  Interventions: Other: Full-fat diet; Other: Low-fat diet
- Low-fat diet first then Full-fat diet (Experimental)
  Interventions: Other: Full-fat diet; Other: Low-fat diet

INTERVENTIONS:
Other: Full-fat diet — The patients will follow a full-fat, isoenergetic diet consisting of 45% carbohydrates, 20% protein, and 35% fat for a duration of three weeks.
Other: Low-fat diet — The patients will follow a low-fat, isoenergetic diet consisting of 45% carbohydrates, 20% protein, and 35% fat for a duration of three weeks.

SUMMARY:
The primary purpose of this study is to determine the impact of whole-fat dairy consumption on cardiovascular and metabolic risk factors and peripheral vascular function in adults with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria: Presence of 3 of the following risk factors:

1. fasting plasma glucose ≥100 mg/dL (or medical therapy for elevated glucose)
2. HDL-C <40 mg/dL in men or <50 mg/dL in women (or medical therapy for reduced HDL-C)
3. Triglycerides ≥150 mg/dL (or medical therapy for elevated triglycerides)
4. Waist circumference >102 cm for men and >88 cm for women
5. Systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥80 mmHg (or medical therapy for hypertension)

Exclusion Criteria:

1. Cardiovascular disease diagnosis
2. Type 1 or 2 diabetes diagnosis
3. Dairy allergy or lactose intolerance
4. Self-reported high baseline dairy intake (>3 servings per day)
5. >3 hours of physical activity per week
6. Pregnant women
7. Inflammatory bowel disease
8. Chronic steroid use
9. Allergy to metal
10. GLP-1 agonist use
11. Patients on medications related to metabolic syndrome where dose adjustments are planned to be made during the study period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change in Total Cholesterol | Baseline, Week 3, Week 5, Week 8
  Total Cholesterol will be measured by a blood sample and reported as mg/dL
Change in HDL-C (High Density Lipoprotein Cholesterol) | Baseline, Week 3, Week 5, Week 8
  High Density Lipoprotein Cholesterol will be measured by a blood sample and reported as mg/dL
Change in LDL-C (Low Density Lipoprotein Cholesterol) | Baseline, Week 3, Week 5, Week 8
  Low Density Lipoprotein Cholesterol will be measured by a blood sample and reported as mg/dL
Change in Triglycerides | Baseline, Week 3, Week 5, Week 8
  Triglycerides will be measured by a blood sample and reported as mg/dL
Change in Blood Glucose | Baseline, Week 3, Week 5, Week 8
  Blood Glucose will be measured by a blood sample and reported as mg/dL
Change in Hemoglobin A1c | Baseline, Week 3, Week 5, Week 8
  Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An A1C level below 5.7 percent is considered normal. Reported as percentage of glycated hemoglobin.
Change in C-reactive protein | Baseline, Week 3, Week 5, Week 8
  C-reactive protein will be measured by a blood sample and reported as mg/L
Change in Lipoprotein | Baseline, Week 3, Week 5, Week 8
  Lipoprotein will be measured by a blood sample and reported as mg/dL
Change in Macrovascular Function | Baseline, Week 3, Week 5, Week 8
  Peripheral macrovascular function is the maximal percent change in brachial artery following cuff release and will be assessed via flow-mediated dilation and reported as a percentage
Change in Microvascular Function | Baseline, Week 3, Week 5, Week 8
  Quantification of the area under the curve of the brachial artery blood flow following cuff release

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Smith, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No